CLINICAL TRIAL: NCT02641704
Title: A Descriptive Study of Characteristics and Progression of Citizens Assigned to a Multidisciplinary Program Focusing on Moving Citizens From Unemployment and Social Security Benefits to Employment and Education
Brief Title: The Development Path
Status: Completed | Type: Observational
Sponsor: University of Southern Denmark (Other)
Collaborators: Sonderborg Municipality (Unknown)
Responsible Party: Principal Investigator, Lotte Nygaard Andersen, Assistant Professor, University of Southern Denmark
Other Study IDs: 14111-SDUpro
Record Dates: First submitted 2015-12-22; First posted 2015-12-29 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Absenteeism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Multidisciplinary program: Multidisciplinary program designed and administered by the Competence- and Integration Center in Sonderborg Municipality
  Interventions: Behavioral: Multidisciplinary program

INTERVENTIONS:
Behavioral: Multidisciplinary program — Coordinated multidisciplinary program

SUMMARY:
The aim of this project is a research-based evaluation of a multidisciplinary program focusing on moving citizens from unemployment and social security benefits to employment and education in Sonderborg Municipality. The citizens who are assigned cannot readily enter the labor market or can get education through employment initiatives in the Job Centre in Sonderborg Municipality because of complex health-related troubles.

The project is designed to include a prospective observational study and a qualitative study using questionnaires, observations, interviews and informations about employment from the Sonderborg Municipality.

ELIGIBILITY:
Inclusion Criteria:

* Assigned to a multidisciplinary program in Sonderborg Municipality (the Law on Active Employment §68 https://www.retsinformation.dk/forms/r0710.aspx?id=164698#Kap2 )

Exclusion Criteria:

* Not able to communicate in Danish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Unemployed citizens with complex health-related problems assigned to a multidisciplinary program in Sønderborg Municipality
Sampling Method: Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Well-being | 12 months
  World Health Organization-5

SECONDARY OUTCOMES:
Well-being | 24 months
  World Health Organization-5
Work ability | 12 months
  10-points Likert scale
Work ability | 24 months
  10-points Likert scale
Pain | 12 months
  Visual analogue scale
Pain | 24 months
  Visual analogue scale
Interpersonal Problems | 12 months
  Inventory of Interpersonal Problems-64
Interpersonal Problems | 24 months
  Inventory of Interpersonal Problems-64
Physical capacity | 12 months
  10-points Likert scale, 5 domains
Physical capacity | 24 months
  10-points Likert scale, 5 domains
Kinesiophobia | 12 months
  Tampa Scale for Kinesiophobia
Kinesiophobia | 24 months
  Tampa Scale for Kinesiophobia
Self-efficacy | 12 months
  General Self-efficacy Scale
Self-efficacy | 24 months
  General Self-efficacy Scale
Depression and anxiety | 12 months
  Patient Health Questionnaire-4
Depression and anxiety | 24 months
  Patient Health Questionnaire-4
Loneliness | 12 months
  Three-item Loneliness Scale
Loneliness | 24 months
  Three-item Loneliness Scale
Ability to work | 12 months
  Registerbased
Ability to work | 24 months
  Registerbased

CONTACTS AND LOCATIONS:
Overall Officials: Lotte Nygaard Andersen, PhD, Principal Investigator — University of Southern Denmark
Locations (1):
- Sønderborg Municipality, Sønderborg, Denmark

REFERENCES:
- [Derived] Andersen LN, Stochkendahl MJ, Roessler KK. En route to flourishing - a longitudinal mixed methods study of long-term unemployed citizens in an interdisciplinary rehabilitation program. BMC Public Health. 2022 Apr 7;22(1):675. doi: 10.1186/s12889-022-13060-9. PMID 35392873
- [Derived] Andersen LN, Stochkendahl MJ, Roessler KK. Parked on the verge: vocational rehabilitation of long-term unemployed citizens - a mixed methods study. Arch Public Health. 2022 Mar 7;80(1):73. doi: 10.1186/s13690-022-00838-x. PMID 35255976
- [Derived] Andersen LN, Stochkendahl MJ, Roessler KK. A municipality-based vocational rehabilitation programme for occupationally marginalized citizens: a study protocol for a mixed methods study. BMC Health Serv Res. 2018 Jul 3;18(1):517. doi: 10.1186/s12913-018-3322-4. PMID 29970107